CLINICAL TRIAL: NCT05445479
Title: Retrospective Study to Identify Whether Doxycycline in SARS-CoV-2 Infection Protects Against Progression to a Severe Form.
Brief Title: Retrospective Study for Identificatiopn of a Link Between Doxycycline and COVID-19 Treatment
Acronym: DOXY-COVID
Status: Withdrawn | Type: Observational
Why Stopped: Study Never Initiated
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_BD_001
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: COVID-19; Doxycycline; Treatment
MeSH Terms: conditions — COVID-19 | interventions — Doxycycline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Doxycycline — Patient with doxycycline treatment during COVID-19 waves

SUMMARY:
A new coronavirus, the third documented animal-to-human passage, emerged in Wuhan , China in the last quarter of 2019. Acne patients on doxycycline escaped seasonal viruses, showing the interest of this antibiotic as a possible treatment against COVID-19.

The antiviral action of tetracyclines can be explained by different mechanisms. First of all, tetracyclines are modulators of innate immunity by decreasing NF-B expression, inhibiting inflammatory cytokines such as TNF-α, IL-1β and IL-6, inflammatory granulomas and free radical release . This action is obtained at doses lower than those necessary to obtain an antibiotic effect. Another possible action of tetracyclines is their ability to chelate zinc from matrix metalloproteinases (MMPS). The coronavirus family is known to bind to host MMPs, particularly for viral survival. Their chelating activity may help inhibit SARS-CoV-2 infection by limiting its ability to replicate in the host. Finally, tetracyclines could have a direct action by inhibiting the replication of single-stranded RNA virus, such as the SARS-CoV-2 coronavirus.We therefore propose a larger comparative study using data from the French National Health Data System.

DETAILED DESCRIPTION:
DOXY-COVID study is a national, observational, retrospective cohort study to compare the risk of severe COVID-19 in doxycycline-treated patients versus non-doxycycline-treated control patients (so-called case-cohort study).

The patient inclusion period corresponds to the main waves associated with the COVID-19 epidemic in France, i.e. from January 1, 2020 to November 30, 2021. Indeed, the time of data access, expected during 2022, would not allow reasonable follow-up of doxycycline-exposed patients from December 1, 2021.

Data of interest collected on these patients are requested over the period from January 1, 2016, through December 31, 2021:

* From January 1, 2016, in order to be able to define a pre-exposure phenotype over a follow-up period of at least 4 years in the French Health Insurance databases (period 2016-2019 inclusive)
* Until December 31, 2021, in order to have at least one month's hindsight on the risk of occurrence of severe forms of COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 12 years old
* Affiliated with the French social security system or equivalent system
* Having been dispensed oral doxycycline at a dose of 100 mg between January 1, 2020 and November 30, 2021

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases are patients with data in the Medicare databases for whom at least one dispensing of doxycycline is identified during the period from January 1, 2020, to December 1, 2021.
  Patients included as cases are all patients identified in the Assurance Maladie databases as having been reimbursed for at least one oral doxycycline dosage form during the period of interest.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of hospitalization associated with COVID-19 | January 1, 2020 to November 30, 2021

IPD SHARING:
Plan to Share IPD: No